CLINICAL TRIAL: NCT04817852
Title: Influence Of Age And Radiograph Presentation on C-Shaped Canal Morphology In Mandibular Second Molar By Using CBCT Analysis
Brief Title: Morphological Root Canal Variation in C-shaped Canal Will be Assessed for Age by Using Cone Beam Computed Tomography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSI College of Dental Sciences and Research, Madurai (Other)
Responsible Party: Principal Investigator, V JASMIN SHAMILI, Principal Investigator, CSI College of Dental Sciences and Research, Madurai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSI
Record Dates: First submitted 2021-03-18; First posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Decayed Teeth
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBCT data of C-shaped canal in mandibular second molar will Be assessed for age. (Experimental): Detection of variation in root canal morphology by using CBCT.
  Interventions: Other: CBCT data of c-shaped canal in mandibular second molar.

INTERVENTIONS:
Other: CBCT data of c-shaped canal in mandibular second molar. — Detection of variation in root canal morphology in mandibular second molar by using CBCT.

SUMMARY:
CBCT Data Of C-Shaped Canal In Mandibular Second Molar Will Be Assessed For Age.

DETAILED DESCRIPTION:
AIM: To determine the influence of age and radiograph presentation on C-shaped canal morphology in mandibular second molar by using CBCT Analysis.

MATERIALS AND METHODS: After obtaining institutional ethics committee approval CSICDSR/IEC/0054/2018 a total of 112 cone beam computed tomography (CBCT) scans from mandibular second molar teeth with C-shaped canal was included for evaluation. These scans were obtained from patients referred to author's department for root canal treatment in the period from July 2016 to March 2020. Informed consent was obtained prior to CBCT scan recommendation. Mandibular molars in this study did not have any root fillings, had fully formed root apices and lack of root resorption. Mandibular second molars in this study were recommended for single tooth CBCT recordings when there was an indication of fused roots in the pre-operative periapical radiograph, with a confirmed C-shaped canal anatomy upon access and / or canal exploration; or with a master cone verification cone shift technique radiograph that a C-shaped canal was evident.

Periapical radiographs were taken with paralleling cone technique using Blue dent X-ray machine (60-70 Kvp, 4-7 mA) and image acquisition was done with Vista Scan Mini plus . The CBCT machine Kodak CS 8100 3D was used for image acquisition with an exposure of 80 KV, 5mA , 19.96 secs and had a voxel size of 90 micro m. All images used 1mm slice thickness.

Periapical radiograph image, axial, coronal and sagittal cross sections of root canal from CBCT were displayed in a monitor and inspected by two experienced endodontic post graduates. Cross sections of root canal were classified according to Fan et al. categorization. Intra- and Inter-observer calibrations had previously been done by assessing 20 selected CBCT volume recording of C-shaped mandibular second molar canal. Two observers analyzed the selected CBCT recordings twice with a 1 week interval between the assessments. Kappa test was done to evaluate the reliability of the observers. The kappa values ranged from 1.000 to 0.761 for inter-and intra-observation reflecting a high level of agreement. Cross section CBCT images were captured

1mm from root canal orifices, at the apical exit of canal and mid-way between the coronal and apical extent of the canal. Any controversies in assessment of images were discussed among the two observers; if consensus was not achieved an experienced endodontic teacher would assist in decision making along with re-examining and scrolling through of CBCT volume recording of the patient in all three planes using the software tools. The periapical radiographs were assessed by an experienced endodontist under 2.5X magnification and optimal light conditions. The C-shaped root appearance in the radiographs was categorized with a modified Gao et al. classification. The modification for the classification was, Type I - Merging: Canals merged into one major canal before exiting at the apical foramen.

Type II - Symmetric: Separated mesial canal and distal canal located at the mesial part and distal part of the root, respectively. Maximum separation between the root canals should be > 1/3rd of distance between the mesial and distal maximum contour of the roots. From the buccal-lingual view, symmetry of the mesial canal and distal canal was present along the longitudinal axis of the root.

Type III - Asymmetric: Separate mesial and distal canals were evident. From a buccal-lingual view, the distal canal may have a large isthmus across the furcation area, which commonly made the mesial and distal canal asymmetrical.

Type IV - Merging symmetric: Canals merged into one major apical exit with partial dentin fusion area may appear in the coronal and (or) middle portion of the canal system. Maximum separation between the root canals should be > 1/3rd of distance between the mesial and distal maximum contour of the roots. Separated mesial and distal canals symmetry was present along the longitudinal axis of the root.

Type V - Merging asymmetric: Canals merged into one major apical exit with partial dentin fusion area may appear in the coronal and (or) middle portion of the canal system. Separated mesial and distal canals asymmetry was present along the longitudinal axis of the root because of presence of large isthmus across the furcation area.

Any variation that could not be accommodated within these established criteria were allocated as variable. C-shaped canal systems in mandibular second molars required three criteria (i) fused roots (ii) a longitudinal groove on the buccal or lingual surface, and (iii) at least one cross section of the canal belonging to classification C1, C2, C3 or C4.

Differences in prevalence of different types of C-shaped root canal configurations between ages were compared using chi-squared test and ANOVA. Statistical analysis was performed using SPSS. P value < 0.05 was considered as significant difference.

ELIGIBILITY:
Inclusion Criteria:

* In lower second molar with C-shaped canal.

Exclusion Criteria:

* Patient not willing for CBCT.

Ages: 13 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Morphological variation in root canal anatomy of c shaped canal in mandibular second molar will be assessed for 180 participants by using cone beam computed tomography | Evaluation of CBCT data up to 2 years.
  To classify the C-shaped canal according to morphology in mandibular second molar by using cone beam computed tomography

SECONDARY OUTCOMES:
Morphological root canal variation in c shaped canal in mandibular second molar will be assessed for 180 participants by using cone beam computed tomography. | Evaluation of CBCT data up to 2 years.
  By using artificial intelligence in detecting c-shaped canal morphology in mandibular second molar.

CONTACTS AND LOCATIONS:
Locations (1):
- CSI College of Dental Sciences And Research, Madurai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No